CLINICAL TRIAL: NCT03282448
Title: Integrated Video-based Family Therapy for Peripartum Depression in Home Visited Mothers: A Pilot Study
Brief Title: Video-based Family Therapy for Peripartum Depression in Home Visited Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fallon P. Cluxton-Keller (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor-Investigator, Fallon P. Cluxton-Keller, Assistant Professor Psychiatry, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 29987; UL1TR001086 (NIH)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Peripartum Depression
MeSH Terms: interventions — Family Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family therapy (Experimental): Adolescent mothers and their family members will receive a total of 10 weekly, 30-minute, video-based family therapy sessions.
  Interventions: Behavioral: family therapy
- Historical comparison group (No Intervention): The Edinburgh Postnatal Depression Scale scores of adolescent mothers in the intervention group will be compared to those of adolescent mothers, who were previously enrolled in the home visiting programs, at the same time points.

INTERVENTIONS:
Behavioral: family therapy — The family-based intervention is informed by Dialectical Behavior Therapy Skills Training for Adolescents (Rathus & Miller, 2014).
  Arms: Family therapy

SUMMARY:
This pilot study will explore the feasibility and acceptability of implementing a family-based treatment, using HIPAA-compliant video-based communication technology, for adolescents (pregnant and post-delivery) with peripartum depressive symptoms within the context of home visiting.

DETAILED DESCRIPTION:
The purpose of the pilot study is to partner with two Federal Maternal, Infant and Early Childhood Home Visiting (HV) Program sites to implement a family-based treatment for depression, using HIPAA-compliant video-based communication technology, in adolescent mothers (pregnant and post-delivery). This implementation-effectiveness hybrid trial includes depressed adolescent mothers and their adult family members.

It has three aims:

1. Explore the feasibility of integrating the treatment model into two Federal HV Program sites in New Hampshire.
2. Test the acceptability of the treatment model among depressed adolescent mothers and their families.
3. Explore preliminary impacts of the treatment on maternal depressive symptoms and parenting attitudes, family emotion regulation, and family functioning at two months post-intervention.

ELIGIBILITY:
Home Visitor Inclusion Criteria:

1. Willingness to participate in the study;
2. Intention to remain in current job for at least 12 months; and
3. Fluency in English: The training, treatment model, implementation meetings, and supervision sessions will be carried out in English.

Family Inclusion Criteria:

1. Adolescent mothers, ages 13-25, in the first trimester of pregnancy through eighteen months postpartum;
2. Adolescent mothers with Edinburgh Postnatal Depression Scale scores of ≥8;
3. At least one of the adolescent mother's family members ("family member" is defined as a person she is biologically related to, or significant close others/partners with whom she is not biologically related) must be willing and available to participate in eight of the 10 video-based family therapy sessions;
4. Fluency in English: The treatment will be carried out in English; and
5. Consistent internet access (i.e., subscribe to an internet service provider and do not experience weekly disruptions in service) on a cell phone, tablet, or computer equipped with a camera and microphone.

Family Exclusion Criteria:

Adolescent mothers with

1. A current positive screen for problem alcohol use on the CAGE or TWEAK;
2. A current positive screen on the drug abuse items on the home visiting interview;
3. A current positive screen for domestic violence on the Relationship Assessment Tool;
4. Current hallucinations and/or delusions;
5. Current homicidal ideation;
6. Current suicidal ideation;
7. Current severe major depressive episode as measured by the SCID-V Depression Module for those over age 18, or NIMH DISC-Y & DISC-P Mood Module for those under age 18; and/or
8. Current self-injurious behavior (e.g., cutting arms on a weekly basis). Families with
9. Current Child Protection Service involvement;
10. Current family therapy service involvement; and/or
11. Current or previous Dialectical Behavior Therapy (DBT) treatment.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Maternal depressive symptoms | 5 months
  Depressive symptoms will be measured using the Beck Depression Inventory (BDI-II; Beck, Steer, & Brown, 1996)

SECONDARY OUTCOMES:
Therapist-family working alliance | 2.5 months
  Clinician rated, and maternal report and family member report.
Family Satisfaction | 2.5 months
  Maternal report and family member report.
Parenting attitudes | 5 months
  A reliable and valid self-report measure will be completed by mothers.
Emotion regulation | 5 months
  A reliable and valid self-report measure will be completed by mothers and their family members.
Family functioning | 5 months
  A reliable and valid self-report measure will be completed by mothers and their family members.

CONTACTS AND LOCATIONS:
Overall Officials: Fallon P. Cluxton-Keller, Ph.D., Principal Investigator — Dartmouth College; Craig L. Donnelly, M.D., Principal Investigator — Dartmouth College; Martha L. Bruce, Ph.D., Study Chair — Dartmouth College
Locations (2):
- United States (2):
  - TLC Family Resource Center, Claremont, New Hampshire
  - The Family Resource Center at Gorham, Gorham, New Hampshire

REFERENCES:
- [Derived] Cluxton-Keller F, Donnelly CL, Williams M, Buteau J, Stolte P, Monroe-Cassel M, Bruce ML. An implementation-effectiveness hybrid trial of video-based family therapy for peripartum depression in home visited mothers: a protocol for a pilot trial. Pilot Feasibility Stud. 2017 Nov 13;3:55. doi: 10.1186/s40814-017-0203-2. eCollection 2017. PMID 29158913